CLINICAL TRIAL: NCT01260350
Title: A Multi-center, Open-Labeled Exploratory Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Oral Administration of PSI-7977 400 mg and Ribavirin for 12 Weeks With and Without Pegylated Interferon in Treatment-Naïve Patients With Chronic HCV Infection Genotype 2 or Genotype 3
Brief Title: Open-Labeled Study of PSI-7977 and RBV With and Without PEG-IFN in Treatment-Naïve Patients With HCV GT2 or GT3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P7977-0523; Medsafe (Other: Medsafe TT50-8648 (1133))
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Hepatitis C Infection
Keywords: PSI-7977; Sofosbuvir; GS-7977; GS-5885; GS-9669; FDC; ribavirin; RBV; Pegylated Interferon; PEG-IFN; Chronic Hepatitis C Infection; HCV; Hepatitis; Genotype 1; Genotype 2; Genotype 3; GT 1; GT 2; GT 3; Hemophilia
MeSH Terms: conditions — Hepatitis; Hemophilia A | interventions — Sofosbuvir; Ribavirin; peginterferon alfa-2a; ledipasvir; GS-9669; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (22):
- Group 1: SOF+RBV 12 wk: GT 2 or 3, TN (Experimental): Treatment-naive (TN) participants with genotype (GT) 2 or 3 HCV infection will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- Group 2: SOF+RBV 12 wk+PEG 4 wk: GT 2 or 3, TN (Experimental): Treatment-naive participants with genotype 2 or 3 HCV infection will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks plus PEG 180 µg once weekly for 4 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: PEG
- Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN (Experimental): Treatment-naive participants with genotype 2 or 3 HCV infection will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks plus PEG 180 µg once weekly for 8 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: PEG
- Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN (Experimental): Treatment-naive participants with genotype 2 or 3 HCV infection will receive SOF 400 mg once daily+weight-based RBV (1000-1200 in a divided daily dose) plus PEG 180 µg once weekly for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: PEG
- Group 5: SOF 12 wk: GT 2 or 3, TN (Experimental): Treatment-naive participants with genotype 2 or 3 HCV infection will receive SOF 400 mg once daily for 12 weeks.
  Interventions: Drug: SOF
- Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN (Experimental): Treatment-naive participants with genotype 2 or 3 HCV infection will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus PEG 180 µg once weekly for 8 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: PEG
- Group 7: SOF+RBV 12 wk: GT 1, TE (Experimental): Treatment-experienced (TE) participants with genotype 1 HCV infection who did not respond to prior treatment will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- Group 8: SOF+RBV 12 wk: GT 1, TN (Experimental): Treatment-naive participants with genotype 1 HCV infection will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- Group 9: SOF+RBV 12 wk: GT 2 or 3, TE (Experimental): Treatment-experienced participants with genotype 2 or 3 HCV infection will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- Group 10: SOF+RBV 8 wk: GT 2 or 3, TN (Experimental): Treatment-naive participants with genotype 2 or 3 HCV infection will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 8 weeks.
  Interventions: Drug: SOF; Drug: RBV
- Group 11: SOF+RBV 12 wk: GT 2 or 3, TN (Experimental): Treatment-naive participants with genotype 2 or 3 HCV infection will receive SOF 400 mg once daily plus split-dose RBV (800 mg in a divided daily dose) for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- Group 12: SOF+RBV+LDV 12 wk: GT 1, TE (Experimental): Treatment-experienced participants with genotype 1 HCV infection who did not respond to prior treatment will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus LDV 90 mg once daily for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: LDV
- Group 13: SOF+RBV+LDV 12 wk: GT 1, TN (Experimental): Treatment-naive participants with genotype 1 HCV infection will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus LDV 90 mg once daily for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: LDV
- Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE (Experimental): Treatment-experienced participants with genotype 1 HCV infection who did not respond to prior treatment will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus GS-9669 500 mg once daily for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: GS-9669
- Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN (Experimental): Treatment-naive participants with genotype 1 HCV infection will receive SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus GS-9669 500 mg once daily for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: GS-9669
- Group 16: LDV/SOF FDC 12 wk: GT 1, fibrosis (Experimental): Treatment-experienced participants with genotype 1 HCV infection and Stage F4 fibrosis who did not respond to prior treatment will receive LDV 90 mg/SOF 400 mg FDC once daily for 12 weeks.
  Interventions: Drug: LDV/SOF
- Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, fibrosis (Experimental): Treatment-experienced participants with genotype 1 HCV infection with Stage F4 fibrosis who did not respond to prior treatment will receive LDV 90 mg/SOF 400 mg FDC once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks.
  Interventions: Drug: RBV; Drug: LDV/SOF
- Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN (Experimental): Treatment-naive participants with genotype 2 or 3 HCV infection will receive LDV 90 mg/SOF 400 mg FDC once daily for 12 weeks.
  Interventions: Drug: LDV/SOF
- Group 19: LDV/SOF FDC 12 wk: GT 2 or 3, TE (Experimental): Treatment-experienced participants with genotype 2 or 3 HCV infection will receive LDV 90 mg/SOF 400 mg FDC once daily for 12 weeks.
  Interventions: Drug: LDV/SOF
- Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, hemophiliac (Experimental): Hemophiliac participants with genotype 1 HCV infection will receive LDV 90 mg/SOF 400 mg FDC once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks.
  Interventions: Drug: RBV; Drug: LDV/SOF
- Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN (Experimental): Treatment-naive participants with genotype 1 HCV infection will receive LDV 90 mg/SOF 400 mg FDC once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 6 weeks.
  Interventions: Drug: RBV; Drug: LDV/SOF
- Group 22: LDV/SOF FDC 6 wk: GT 1, TN (Experimental): Treatment-naive participants with genotype 1 HCV infection were randomized to receive LDV 90 mg/SOF 400 mg FDC once daily for 6 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) tablets administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Arms: Group 10: SOF+RBV 8 wk: GT 2 or 3, TN; Group 11: SOF+RBV 12 wk: GT 2 or 3, TN; Group 12: SOF+RBV+LDV 12 wk: GT 1, TE; Group 13: SOF+RBV+LDV 12 wk: GT 1, TN; Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE; Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN; Group 1: SOF+RBV 12 wk: GT 2 or 3, TN; Group 2: SOF+RBV 12 wk+PEG 4 wk: GT 2 or 3, TN; Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN; Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN; Group 5: SOF 12 wk: GT 2 or 3, TN; Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN; Group 7: SOF+RBV 12 wk: GT 1, TE; Group 8: SOF+RBV 12 wk: GT 1, TN; Group 9: SOF+RBV 12 wk: GT 2 or 3, TE
Drug: RBV — Ribavirin (RBV) capsules administered orally in a divided daily dose
  Other Names: Copegus®
  Arms: Group 10: SOF+RBV 8 wk: GT 2 or 3, TN; Group 11: SOF+RBV 12 wk: GT 2 or 3, TN; Group 12: SOF+RBV+LDV 12 wk: GT 1, TE; Group 13: SOF+RBV+LDV 12 wk: GT 1, TN; Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE; Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN; Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, fibrosis; Group 1: SOF+RBV 12 wk: GT 2 or 3, TN; Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, hemophiliac; Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN; Group 2: SOF+RBV 12 wk+PEG 4 wk: GT 2 or 3, TN; Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN; Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN; Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN; Group 7: SOF+RBV 12 wk: GT 1, TE; Group 8: SOF+RBV 12 wk: GT 1, TN; Group 9: SOF+RBV 12 wk: GT 2 or 3, TE
Drug: PEG — Peginterferon alfa-2a (PEG) administered via subcutaneous injection once weekly
  Other Names: Pegasys®
  Arms: Group 2: SOF+RBV 12 wk+PEG 4 wk: GT 2 or 3, TN; Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN; Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN; Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN
Drug: LDV — Ledipasvir (LDV) tablets administered orally once daily
  Other Names: GS-5885
  Arms: Group 12: SOF+RBV+LDV 12 wk: GT 1, TE; Group 13: SOF+RBV+LDV 12 wk: GT 1, TN
Drug: GS-9669 — GS-9669 tablets administered orally once daily
  Arms: Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE; Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN
Drug: LDV/SOF — LDV/SOF fixed-dose combination (FDC) tablet administered once daily
  Other Names: Harvoni®
  Arms: Group 16: LDV/SOF FDC 12 wk: GT 1, fibrosis; Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, fibrosis; Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN; Group 19: LDV/SOF FDC 12 wk: GT 2 or 3, TE; Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, hemophiliac; Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN; Group 22: LDV/SOF FDC 6 wk: GT 1, TN

SUMMARY:
This study is to assess the safety and tolerability of sofosbuvir (SOF) 400 mg with and without ribavirin (RBV) and/or with and without pegylated interferon alfa-2a (PEG) in subjects with genotype 1, 2 or 3 hepatitis C (HCV) infection.

DETAILED DESCRIPTION:
Part 1: HCV genotype 2 or 3: participants will receive SOF 400 mg once daily with weight-based RBV for 12 weeks. Participants will be randomized in equal proportions to: no PEG (Arm 1), PEG for 4 weeks (Arm 2), PEG for 8 weeks (Arm 3), or PEG for 12 weeks (Arm 4).

Part 2: HCV genotype 2 or 3: participants will receive SOF 400 mg once daily (monotherapy) for 12 weeks (Arm 5), or SOF 400 mg once daily with PEG and weight-based RBV for 8 weeks (Arm 6); HCV genotype 1: null responders (did not respond to their prior treatment) will receive SOF 400 mg once daily with weight-based RBV for 12 weeks (Arm 7).

Part 3: HCV genotype 1 treatment-naive (Arm 8) or HCV genotype 2 or 3 treatment-experienced participants (Arm 9) will receive SOF 400 mg once daily in combination with weight-based RBV for 12 weeks.

Part 4: HCV genotype 2 or 3 treatment naive participants will receive SOF 400 mg once daily with weight-based RBV for 8 weeks (Arm 10) or SOF 400 mg once daily and 800 mg RBV for 12 weeks (Arm 11). HCV genotype 1 null responders will receive SOF 400 mg once daily, ledipasvir (LDV), and weight based RBV for 12 weeks (Arm 12). HCV genotype-1 treatment naive participants will receive SOF 400 mg once daily with weight-based RBV and LDV for 12 weeks (Arm 13).

Part 5: HCV genotype 1 null responders will receive SOF 400 mg once daily with GS-9669 500 mg once daily and weight-based RBV for 12 weeks (Arm 14). HCV genotype-1 treatment naive participants receive SOF 400 mg once daily with GS-9669 500 mg once daily and weight-based RBV for 12 weeks (Arm 15).

Part 6: HCV genotype 1 null responders with Stage F4 fibrosis will receive LDV/SOF FDC for 12 weeks (Arm 16) or LDV/SOF FDC with weight-based RBV for 12 weeks (Arm 17). HCV genotype 2 or 3 treatment-naive participants will receive LDV/SOF FDC for 12 weeks (Arm 18). HCV genotype 2 or 3 treatment-experienced participants will receive LDV/SOF FDC for 12 weeks (Arm 19). HCV genotype 1 hemophiliacs will receive LDV/SOF FDC with weight-based RBV for 12 weeks (Arm 20). HCV genotype 1 treatment-naive participants will receive LDV/SOF FDC with weight-based RBV for 6 weeks (Arm 21). HCV genotype 1 treatment-naive participants will receive LDV/SOF FDC for 6 weeks (Arm 22).

ELIGIBILITY:
Inclusion Criteria:

* Chronic Genotype 2 or 3 HCV-infection or Genotype 1, serum HCV RNA ≥ 50,000 IU/mL
* Not co-infected with HIV
* Use of highly effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* History of any other clinically significant chronic liver disease
* Pregnant or nursing female or male with pregnant female partner
* History of significant drug allergy to nucleoside/nucleotide analogs.
* Participation in a clinical study within 3 months prior to first dose
* Positive result for significant drug use at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2010-12; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Hyland, DPhil, Study Director — Gilead Sciences
Locations (2):
- New Zealand (2):
  - Auckland Clinical Studies Ltd., Auckland
  - Christchurch Clinical Studies Trust, Christchurch

REFERENCES:
- [Result] Gane EJ, Stedman CA, Hyland RH, Ding X, Svarovskaia E, Subramanian GM, Symonds WT, McHutchison JG, Pang PS. Efficacy of nucleotide polymerase inhibitor sofosbuvir plus the NS5A inhibitor ledipasvir or the NS5B non-nucleoside inhibitor GS-9669 against HCV genotype 1 infection. Gastroenterology. 2014 Mar;146(3):736-743.e1. doi: 10.1053/j.gastro.2013.11.007. Epub 2013 Nov 18. PMID 24262278
- [Result] Gane EJ, Stedman CA, Hyland RH, Ding X, Svarovskaia E, Symonds WT, Hindes RG, Berrey MM. Nucleotide polymerase inhibitor sofosbuvir plus ribavirin for hepatitis C. N Engl J Med. 2013 Jan 3;368(1):34-44. doi: 10.1056/NEJMoa1208953. PMID 23281974

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in a total of 2 study sites in New Zealand. The first participant was screened on 18 November 2010. The last participant observation was on 23 December 2013.
Groups:
- Group 1: SOF+RBV 12 wk: GT 2 or 3, TN: Sofosbuvir (SOF) 400 mg once daily plus weight-based ribavirin (RBV) (1000-1200 in a divided daily dose) for 12 weeks in treatment-naive (TN) participants with genotype (GT) 2 or 3 HCV infection
- Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks plus PEG 180 µg once weekly for 4 weeks in treatment-naive participants with genotype 2 or 3 HCV infection
- Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks plus PEG 180 µg once weekly for 8 weeks in treatment-naive participants with genotype 2 or 3 HCV infection
- Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus PEG 180 µg once weekly for 12 weeks in treatment-naive participants with genotype 2 or 3 HCV infection
- Group 5: SOF 12 wk: GT 2 or 3, TN: SOF 400 mg once daily for 12 weeks in treatment-naive participants with genotype 2 or 3 HCV infection
- Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus PEG 180 µg once weekly for 8 weeks in treatment-naive participants with genotype 2 or 3 HCV infection
- Group 7: SOF+RBV 12 wk: GT 1, TE: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks in treatment-experienced (TE) participants with genotype 1 HCV infection who did not respond to prior treatment
- Group 8: SOF+RBV 12 wk: GT 1, TN: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks in treatment-naive participants with genotype 1 HCV infection
- Group 9: SOF+RBV 12 wk: GT 2 or 3, TE: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks in treatment-experienced participants with genotype 2 or 3 HCV infection
- Group 10: SOF+RBV 8 wk: GT 2 or 3, TN: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 8 weeks in treatment-naive participants with genotype 2 or 3 HCV infection
- Group 11: SOF+RBV 12 wk: GT 2 or 3, TN: SOF 400 mg once daily plus split-dose RBV (800 mg in a divided daily dose) for 12 weeks in treatment-naive participants with genotype 2 or 3 HCV infection
- Group 12: SOF+RBV+LDV 12 wk: GT 1, TE: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus ledipasvir (LDV) 90 mg once daily for 12 weeks in treatment-experienced participants with genotype 1 HCV infection who did not respond to prior treatment
- Group 13: SOF+RBV+LDV 12 wk: GT 1, TN: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus LDV 90 mg once daily for 12 weeks in treatment-naive participants with genotype 1 HCV infection
- Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus GS-9669 500 mg once daily for 12 weeks in treatment-experienced participants with genotype 1 HCV infection who did not respond to prior treatment
- Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus GS-9669 500 mg once daily for 12 weeks in treatment-naive participants with genotype 1 HCV infection
- Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis: LDV 90 mg/SOF 400 mg fixed-dose combination (FDC) once daily for 12 weeks in treatment-experienced participants with genotype 1 HCV infection with Stage F4 fibrosis who did not respond to prior treatment
- Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis: LDV 90 mg/SOF 400 mg FDC once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks in treatment-experienced participants with genotype 1 HCV infection with Stage F4 fibrosis who did not respond to prior treatment
- Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN: LDV 90 mg/SOF 400 mg FDC once daily for 12 weeks in treatment-naive participants with genotype 2 or 3 HCV infection
- Group 19: LDV/SOF FDC 12 wk: GT 2 or 3, TE: LDV 90 mg/SOF 400 mg FDC once daily for 12 weeks in treatment-experienced participants with genotype 2 or 3 HCV infection
- Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac: LDV 90 mg/SOF 400 mg FDC once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks in hemophiliac participants with genotype 1 HCV infection
- Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN: LDV 90 mg/SOF 400 mg FDC once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 6 weeks in treatment-naive participants with genotype 1 HCV infection
Period: Overall Study
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 19: LDV/SOF FDC 12 wk: GT 2 or 3, TE | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN | Group 22: LDV/SOF FDC 6 wk: GT 1, TN
Started | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 10 | 0 | 14 | 25 | 0
Completed | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 24 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 9 | 0 | 14 | 22 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Not completed — Did Not Complete Follow-up 12 Visit | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least one dose of study medication.
Groups:
- Group 1: SOF+RBV 12 wk: GT 2 or 3, TN: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) for 12 weeks in treatment-naive (TN) participants with genotype (GT) 2 or 3 HCV infection
- Group 12: SOF+RBV+LDV 12 wk: GT 1, TE: SOF 400 mg once daily plus weight-based RBV (1000-1200 in a divided daily dose) plus LDV 90 mg once daily for 12 weeks in treatment-experienced participants with genotype 1 HCV infection who did not respond to prior treatment
- Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis: LDV 90 mg/SOF 400 mg FDC once daily for 12 weeks in treatment-experienced participants with genotype 1 HCV infection with Stage F4 fibrosis who did not respond to prior treatment
- Total: Total of all reporting groups
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN | Total
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 10 | 14 | 25 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (6.0) | 47 (10.2) | 49 (9.9) | 46 (6.3) | 43 (13.5) | 39 (12.2) | 48 (10.4) | 48 (11.4) | 53 (7.9) | 48 (9.4) | 39 (8.9) | 50 (13.0) | 45 (9.2) | 55 (6.0) | 46 (9.3) | 61 (4.9) | 57 (5.2) | 39 (10.8) | 54 (13.0) | 51 (9.0) | 48 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 2 | 6 | 5 | 3 | 10 | 6 | 8 | 3 | 2 | 17 | 3 | 12 | 0 | 1 | 7 | 2 | 12 | 110
  Male | 8 | 5 | 5 | 9 | 4 | 5 | 7 | 15 | 19 | 17 | 7 | 7 | 8 | 7 | 13 | 10 | 8 | 3 | 12 | 13 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 10 | 9 | 10 | 11 | 10 | 9 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 8 | 9 | 10 | 14 | 25 | 289
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7 | 4 | 8 | 9 | 10 | 7 | 9 | 20 | 17 | 20 | 9 | 9 | 23 | 9 | 20 | 8 | 9 | 7 | 12 | 22 | 239
  Asian | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 11
  Native Hawaiian of Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 3 | 4 | 0 | 2 | 0 | 3 | 1 | 3 | 6 | 3 | 0 | 0 | 1 | 1 | 4 | 2 | 0 | 0 | 1 | 2 | 36
Hepatitis C Virus (HCV) RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.7 (0.42) | 6.6 (0.52) | 6.4 (0.57) | 6.3 (0.76) | 5.7 (0.89) | 6.1 (0.88) | 6.8 (0.55) | 6.1 (0.75) | 6.5 (0.66) | 6.1 (0.80) | 6.2 (0.96) | 6.9 (0.20) | 5.9 (0.85) | 7.0 (0.38) | 6.3 (0.54) | 6.5 (0.57) | 6.3 (0.78) | 6.1 (0.94) | 6.5 (0.51) | 6.5 (0.56) | 6.3 (0.73)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 1 | 1 | 3 | 3 | 5 | 5 | 1 | 10 | 5 | 12 | 4 | 0 | 11 | 0 | 8 | 2 | 3 | 5 | 2 | 6 | 87
  ≥ 6 log10 IU/mL | 9 | 8 | 7 | 8 | 5 | 5 | 9 | 15 | 20 | 13 | 6 | 9 | 14 | 10 | 17 | 8 | 6 | 5 | 12 | 19 | 205
HCV Genotype [Number; unit: participants] — There are variations of HCV which are all similar enough to be called HCV, but are distinct enough to be referred to as HCV genotypes.
  participants
    Genotype 1 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 25 | 0 | 0 | 0 | 9 | 25 | 10 | 25 | 10 | 9 | 0 | 14 | 25 | 162
    Genotype 2 | 4 | 3 | 4 | 4 | 3 | 0 | 0 | 0 | 6 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 31
    Genotype 3 | 6 | 6 | 6 | 7 | 7 | 10 | 0 | 0 | 19 | 20 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 99
IL28b Genotype [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 5 | 4 | 4 | 4 | 2 | 3 | 10 | 25 | 0 | 13 | 4 | 0 | 9 | 1 | 7 | 4 | 2 | 3 | 4 | 5 | 109
    CT | 4 | 4 | 4 | 5 | 6 | 6 | 0 | 0 | 6 | 12 | 5 | 7 | 14 | 8 | 14 | 4 | 5 | 6 | 7 | 15 | 132
    TT | 1 | 1 | 2 | 2 | 2 | 1 | 0 | 0 | 19 | 0 | 1 | 2 | 2 | 1 | 4 | 2 | 2 | 1 | 3 | 5 | 51
Cirrhosis Status [Number; unit: participants]
  Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 9 | 0 | 1 | 0 | 20
  No | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 0 | 0 | 10 | 13 | 25 | 272

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Adverse Events
Description: Adverse events (AEs) occurring from baseline (Day 1 for all groups) to 30 days following the last dose of study drug were summarized across the participant population. A participant was counted once if they had a qualifying event.
Time Frame: Up to 12 weeks plus 30 days
Population: Safety Analysis Set: participants were randomized and received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 10 | 14 | 25
Percentage of participants
  Any AE | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 24 | 25 | 10 | 9 | 24 | 10 | 25 | 7 | 8 | 7 | 13 | 22
  Drug-related AE | 8 | 9 | 10 | 11 | 7 | 10 | 10 | 25 | 20 | 21 | 7 | 9 | 24 | 10 | 21 | 5 | 8 | 6 | 12 | 19
  Grade 3 or higher AE | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 0 | 1 | 0
  AE leading to drug discontinuation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2
  Serious AE | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Following Completion of Treatment (SVR12)
Description: SVR12 was defined as HCV RNA < the limit of detection (LOD; < 15 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 10 | 14 | 25
percentage of participants | 100.0 [69.2 to 100.0] | 100.0 [66.4 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [71.5 to 100.0] | 60.0 [26.2 to 87.8] | 100.0 [69.2 to 100.0] | 10.0 [0.3 to 44.5] | 84.0 [63.9 to 9] | 68.0 | 64.0 [42.5 to 82.0] | 60.0 [26.2 to 87.8] | 100.0 [66.4 to 100.0] | 100.0 [86.3 to 100.0] | 100.0 [69.2 to 100.0] | 92.0 [74.0 to 99.0] | 70.0 | 100.0 | 80.0 | 100.0 | 68.0

3. Secondary Outcome: Percentage of Participants With HCV RNA < LOD at Week 6
Time Frame: Week 6
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 10 | 14 | 25
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

4. Secondary Outcome: Percentage of Participants With HCV RNA < LOD at Week 8
Description: Data are not presented for Group 21 which ended treatment after Week 6.
Time Frame: Week 8
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 10 | 14
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

5. Secondary Outcome: Percentage of Participants With HCV RNA < LOD at Week 12
Description: Data are not presented for Groups 6, 10, and 21 which ended treatment after Week 8 or Week 6.
Time Frame: Week 12
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 25 | 25 | 10 | 9 | 24 | 10 | 25 | 10 | 9 | 10 | 14
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

6. Secondary Outcome: Change From Baseline in HCV RNA at Week 6
Time Frame: Baseline to Week 6
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 10 | 14 | 25
log10 IU/mL | -5.52 (0.418) | -5.44 (0.519) | -5.23 (0.571) | -5.20 (0.756) | -6.23 (0.892) | -4.94 (0.885) | -5.70 (0.550) | -4.95 (0.746) | -5.38 (0.660) | -4.92 (0.803) | -5.01 (0.962) | -5.74 (0.203) | -4.80 (0.851) | -5.84 (0.383) | -5.19 (0.536) | -5.36 (0.575) | -5.18 (0.781) | -4.93 (0.942) | -5.35 (0.510) | -5.39 (0.559)

7. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Description: Data are not presented for Group 21 which ended treatment after Week 6.
Time Frame: Baseline to Week 8
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 10 | 14
log10 IU/mL | -5.52 (0.418) | -5.44 (0.519) | -5.23 (0.571) | -5.20 (0.756) | -4.59 (0.892) | -4.94 (0.885) | -5.70 (0.550) | -4.95 (0.746) | -5.38 (0.660) | -4.92 (0.803) | -5.01 (0.962) | -5.74 (0.203) | -4.80 (0.851) | -5.84 (0.383) | -5.19 (0.536) | -5.36 (0.575) | -5.18 (0.781) | -4.93 (0.942) | -5.35 (0.510)

8. Secondary Outcome: Change From Baseline in HCV RNA at Week 12
Description: Data are not presented for Groups 6, 10, and 21 which ended treatment after Week 8 or Week 6. Data are not presented for Groups 16, 17, 18, and 20 because participants with detectable HCV RNA discontinued due to protocol-specified stopping rules.
Time Frame: Baseline to Week 12
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 25 | 25 | 10 | 9 | 24 | 10 | 25
log10 IU/mL | -5.52 (0.418) | -5.44 (0.519) | -5.23 (0.571) | -5.20 (0.756) | -4.59 (0.892) | -5.70 (0.550) | -4.95 (0.746) | -5.39 (0.660) | -2.01 (0.962) | -5.74 (0.203) | -4.85 (0.823) | -5.84 (0.383) | -5.19 (0.536)

9. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: The percentage of participants with on-treatment virologic failure (viral breakthrough, rebound, or nonresponse) or following treatment (viral relapse) was summarized.
  On-treatment virologic failure was defined as:
  * Viral breakthrough (confirmed HCV RNA ≥ LOD after having previously had HCV RNA < LOD while on treatment),
  * Viral rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment, or
  * Nonresponse (HCV RNA persistently ≥ LOD through 6 weeks of treatment)
  Viral relapse was defined as confirmed HCV RNA ≥ LOD during the posttreatment period having achieved HCV RNA < LOD at the last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN
Number analyzed (Participants) | 10 | 9 | 10 | 11 | 10 | 10 | 10 | 25 | 25 | 25 | 10 | 9 | 25 | 10 | 25 | 10 | 9 | 10 | 14 | 25
percentage of participants
  On-treatment virologic failure | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Viral relapse | 0.0 | 0.0 | 0.0 | 0.0 | 40.0 | 0.0 | 90.0 | 16.0 | 32.0 | 36.0 | 40.0 | 0.0 | 0.0 | 0.0 | 8.0 | 30.0 | 0.0 | 20.0 | 0.0 | 32.0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days.
Description: Adverse events are included up to the last dose date of any study drug + 30 days.
Arm/Group | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN | Group 5: SOF 12 wk: GT 2 or 3, TN | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN | Group 7: SOF+RBV 12 wk: GT 1, TE | Group 8: SOF+RBV 12 wk: GT 1, TN | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/9 | 0/10 | 0/11 | 0/10 | 1/10 | 0/10 | 1/25 | 0/25 | 2/25 | 0/10 | 0/9 | 2/25 | 0/10 | 0/25 | 0/10 | 0/9 | 0/10 | 2/14 | 0/25
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9 | 10/10 | 11/11 | 10/10 | 10/10 | 10/10 | 25/25 | 24/25 | 25/25 | 10/10 | 9/9 | 24/25 | 10/10 | 25/25 | 7/10 | 8/9 | 7/10 | 13/14 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN (N=10) | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN (N=9) | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN (N=10) | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN (N=11) | Group 5: SOF 12 wk: GT 2 or 3, TN (N=10) | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN (N=10) | Group 7: SOF+RBV 12 wk: GT 1, TE (N=10) | Group 8: SOF+RBV 12 wk: GT 1, TN (N=25) | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE (N=25) | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN (N=25) | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN (N=10) | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE (N=9) | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN (N=25) | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE (N=10) | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN (N=25) | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis (N=10) | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis (N=9) | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN (N=10) | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac (N=14) | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN (N=25)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Emterovesical Fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: SOF+RBV 12 wk: GT 2 or 3, TN (N=10) | Group 2: SOF+RBV 12 wk +PEG 4 wk: GT 2 or 3, TN (N=9) | Group 3: SOF+RBV 12 wk+PEG 8 wk: GT 2 or 3, TN (N=10) | Group 4: SOF+RBV+PEG 12 wk: GT 2 or 3, TN (N=11) | Group 5: SOF 12 wk: GT 2 or 3, TN (N=10) | Group 6: SOF+RBV+PEG 8 wk: GT 2 or 3, TN (N=10) | Group 7: SOF+RBV 12 wk: GT 1, TE (N=10) | Group 8: SOF+RBV 12 wk: GT 1, TN (N=25) | Group 9: SOF+RBV 12 wk: GT 2 or 3, TE (N=25) | Group 10: SOF+RBV 8 wk: GT 2 or 3, TN (N=25) | Group 11: SOF+RBV 12 wk: GT 2 or 3, TN (N=10) | Group 12: SOF+RBV+LDV 12 wk: GT 1, TE (N=9) | Group 13: SOF+RBV+LDV 12 wk: GT 1, TN (N=25) | Group 14: SOF+RBV+GS-9669 12 wk: GT 1, TE (N=10) | Group 15: SOF+RBV+GS-9669 12 wk: GT 1, TN (N=25) | Group 16: LDV/SOF FDC 12 wk: GT 1, Fibrosis (N=10) | Group 17: LDV/SOF FDC+RBV 12 wk: GT 1, Fibrosis (N=9) | Group 18: LDV/SOF FDC 12 wk: GT 2 or 3, TN (N=10) | Group 20: LDV/SOF FDC+RBV 12 wk: GT 1, Hemophiliac (N=14) | Group 21: LDV/SOF FDC+RBV 6 wk: GT 1, TN (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 5 | 1 | 2 | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pterygium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 2 | 0 | 3 | 1 | 6 | 1 | 3 | 1 | 1 | 2 | 0 | 4 | 0 | 0 | 3 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 4 | 2 | 3 | 2 | 2 | 11 | 5 | 4 | 3 | 3 | 6 | 2 | 9 | 0 | 4 | 1 | 4 | 5
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 9 | 0 | 2 | 1 | 1 | 3
Application site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crying (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 3 | 5 | 3 | 7 | 4 | 12 | 10 | 9 | 1 | 7 | 6 | 5 | 4 | 1 | 1 | 0 | 7 | 6
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 2 | 0 | 1 | 4 | 1 | 2 | 1 | 5 | 0 | 3 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 1 | 2 | 3
Malaise (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 2 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 6 | 3 | 3 | 3 | 9 | 2 | 3 | 1 | 1 | 2 | 2 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3 | 0 | 5 | 0 | 2 | 2 | 3 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1 | 0 | 1 | 1 | 3 | 0 | 2 | 1 | 0 | 5 | 2 | 2 | 0 | 2 | 0 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 3 | 1 | 4 | 0 | 2 | 6 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 4 | 4 | 2 | 3 | 2 | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 7 | 9 | 8 | 8 | 6 | 4 | 8 | 11 | 6 | 2 | 6 | 11 | 4 | 8 | 3 | 2 | 4 | 5 | 8
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 2 | 3 | 4 | 1 | 0 | 0 | 3 | 0 | 1 | 2 | 2 | 0 | 1 | 2
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 4 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Depressive symptom (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphoria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysthymic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impatience (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 6 | 5 | 5 | 6 | 1 | 4 | 5 | 3 | 3 | 2 | 4 | 4 | 1 | 3 | 0 | 1 | 2 | 3 | 6
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Loss of libido (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 3
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 0 | 0 | 2 | 1 | 1 | 4 | 1 | 0 | 1 | 5 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 2 | 0 | 2 | 2 | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 3 | 1 | 6 | 3 | 4 | 6 | 1 | 1 | 1 | 4 | 1 | 5 | 0 | 0 | 1 | 1 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years